CLINICAL TRIAL: NCT05115734
Title: Acylcarnitine Profile After Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, University of Liege
Other Study IDs: CARNUSI
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Critical Care; Carnitine Metabolism Disturbances

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short stayers: Determination of the acylcarnitine profile during the 5 days following discharge of a short stay in ICU (maximum 2 days)
  Interventions: Diagnostic Test: Serum acylcarnitine profiling
- Long stayers: Determination of the acylcarnitine profile during the year following discharge of a prolonged stay in ICU (7 days or more)
  Interventions: Diagnostic Test: Serum acylcarnitine profiling

INTERVENTIONS:
Diagnostic Test: Serum acylcarnitine profiling — Blood samples are collected through a central or peripheral venous line placed for clinical use, or through venous punction. Blood will be drawn into a serum gel tube (BD Vacutainer, Becton, Dickinson and Company, Franklin Lakes, NJ, USA), before being centrifuged (3500 rpm, 15 min, 4°C). Supernatant will be frozen at -20°C and stored for later analysis.
  Serum ACs concentrations (free carnitine (C0), C2-, C3-, C3DC-, C4-, C4-OH-, C4-DC-, C5-, C5:1-, C5-OH-, C5DC-, C6-, C6-OH-, C6-DC-, C8-, C8:1-, C10-, C10:1-, C10:2-, C12-, C12:1-, C14-, C14:1-, C14:2-, C14-OH-, C16-, C16:1-, C16-OH-, C16-1-OH-, C17-, C18- ,C18:1-, C18:2-, C18-OH-, C18:1-OH-, C18:2-OH-carnitine) will be determined on a TQ5500 tandem mass spectrometer (Sciex, Framingham, MA, USA).

SUMMARY:
The aim of the study is to compare the acylcarnitine profile of critically ill survivors of a prolonged stay in ICU with the profile of survivors of short ICU length of stay. The second aim is to assess the evolution of the acylcarnitine profile over time in survivors of a prolonged ICU stay.

DETAILED DESCRIPTION:
In a retrospective analysis focused on survivors of an ICU stay of 7 days or more, we showed that during the week following discharge, carnitine deficiency was rare, but acylcarnitine profile was altered, with an abnormal acylcarnitine/carnitine ratio in more than 25% of the population.

Carnitine has a key role in cellular energy metabolism and is a a biomarker of the mitochondria function. Moreover, mitochondrial function is proven to be severely impaired in critically ill patients and mitochondrial dysfunction has been linked to post-ICU disorders.

In this context, it is relevant to study the evolution over time of the acylcarnitine profile in ICU survivors of a prolonged ICU stay. It is also relevant to compare the same profile between survivors of a prolonged and a shorter ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Group short stayers: ICU length of stay of 2 days
* Group long stayers: ICU length of stay of at least 7 days

Exclusion criteria: patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Group short stayers: Critically ill patients with ICU length of stay of 2 days: patients admitted in ICU after a scheduled cardiac surgery with sternotomy
  * Group long stayers: Critically ill patients with ICU length of stay of at least 7 days, whatever the critically illness
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Acylcarnitine profile | During the 5 first days following ICU discharge
  Serum acylcarnitine profile
Acylcarnitine profile | 1 month following ICU discharge
  Serum acylcarnitine profile in long stayers
Acylcarnitine profile | 3 month following ICU discharge
  Serum acylcarnitine profile in long stayers
Acylcarnitine profile | 12 month following ICU discharge
  Serum acylcarnitine profile in long stayers

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No